CLINICAL TRIAL: NCT07031167
Title: The COMFORTage Project: Integration of Multiple Sources Towards Personalized Preventions at Ace Alzheimer Center Barcelona
Brief Title: The COMFORTage Project at Ace Alzheimer Center Barcelona
Acronym: COMFORTage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació ACE Institut Català de Neurociències Aplicades (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: comfortage_ace_1
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Active Functional Intervention (No Intervention): No stimulation activity
- Active Functional Intervention (Experimental): Stimulation activity
  Interventions: Behavioral: Cognitive and functional stimulation using digital platforms

INTERVENTIONS:
Behavioral: Cognitive and functional stimulation using digital platforms — Participants in the intervention group receive personalized cognitive and functional stimulation over one year through digital platforms developed by the COMFORTage project. These include Eligence, a brain-training tool featuring interactive games targeting memory, attention, and language; Language Games, which assess and train linguistic and cognitive skills in realistic scenarios; and Healthentia, a platform that monitors daily health metrics and provides virtual coaching. Sessions are conducted both in person and remotely, and are adapted to each participant's abilities and level of digital literacy. The intervention aims to support cognitive health and daily functioning in individuals with MCI or mild AD.
  Arms: Active Functional Intervention

SUMMARY:
The COMFORTage study at Ace Alzheimer Center Barcelona is investigating whether a personalized cognitive and functional stimulation program can help slow cognitive decline in individuals diagnosed with mild cognitive impairment (MCI) or mild Alzheimer's disease (AD) dementia.

The study involves 100 participants aged 60 to 85, who are randomly assigned to one of two groups. The active group receives weekly in-person sessions for one year, featuring individualized cognitive and physical training through digital platforms developed by the COMFORTage project. The control group does not participate in the training but undergoes the same schedule of health assessments and monitoring.

All participants are followed for a total of two years. Throughout the study, researchers collect comprehensive clinical, neuropsychological, and biological data. This includes cognitive assessments, magnetic resonance imaging (MRI) brain scans, blood and cerebrospinal fluid (CSF) samples, and genetic testing. In addition, participants complete spontaneous speech recordings from home every 3-4 months using a dedicated mobile application.

The primary objective is to determine whether the stimulation program more effectively preserves memory and cognitive function compared to no intervention. The study also evaluates its impact on physical and emotional well-being, daily functioning, and quality of life. Insights from the trial will contribute to the development of an artificial intelligence (AI)-powered digital health platform aimed at delivering personalized care for individuals living with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 85 years.
* Diagnosis of MCI based on Petersen criteria with a CDR score of 0.5.
* Diagnosis of mild AD dementia according to National Institute on Aging-Alzheimer's Association (NIA-AA) criteria with a CDR score of 1.
* Proficiency in using digital tools such as mobile apps, tablets, or computers.
* Ability and willingness to attend regular in-person sessions at Ace Alzheimer Center Barcelona.
* Provided written informed consent after receiving a full explanation of the study.

Exclusion Criteria:

* History of traumatic brain injury.
* Diagnosis of severe depression.
* History of stroke or brain tumors.
* Presence of significant uncorrected visual or auditory impairments.
* Lack of access to a digital device or internet connection.
* Inability to participate in regular in-person sessions at the study site.
* Any medical condition that may confound cognitive assessment or limit participation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in neuropsychological assessment | Baseline, 1-year follow-up, and 2-year follow-up
  Assesses the change in cognitive function over two years using composite scores from the Neuropsychological Battery used at Ace (NBACE). The scores evaluate five domains: attention, memory, visuospatial/visuoperceptual functions, executive functions, and language. The scores for each domain range from -3 (low competence) to 3 (high competence).

SECONDARY OUTCOMES:
Change in Mini-Mental State Examination (MMSE) score | Baseline, 1-year follow-up, and 2-year follow-up
  This test is administered to assess general cognitive function. Results are expressed as points on a scale from 0 (severe cognitive impairment) to 30 (normal cognitive function).
Change in Memory Test Score from the 7-Minute Screen Test (Spanish version) | Baseline, 1-year follow-up, and 2-year follow-up
  This test measures memory recall for cognitive screening purposes. The unit of measure is points on a scale from 0 (poor recall) to 7 (excellent recall).
Change in Hachinski Ischemia Scale score | Baseline, 1-year follow-up, and 2-year follow-up
  This scale evaluates the vascular contribution to cognitive impairment. Scores range from 0 (pure Alzheimer's disease) to 18 (multi-infarct dementia likely).
Change in Neuropsychiatric Inventory Questionnaire (NPI-Q) score | Baseline, 1-year follow-up, and 2-year follow-up
  NPI-Q assesses behavioral and psychological symptoms in dementia, using a scale from 0 to 36 where higher scores indicate greater symptom severity and caregiver distress.
Change in Global Deterioration Scale (GDS) score | Baseline, 1-year follow-up, and 2-year follow-up
  GDS assesses stages of cognitive decline from normal aging to severe dementia. Scores range from 1 (no cognitive decline) to 7 (very severe cognitive decline).
Change in Clinical Dementia Rating (CDR) score | Baseline, 1-year follow-up, and 2-year follow-up
  CDR evaluates the severity of dementia symptoms across multiple domains, using a global score from 0 (no dementia) to 3 (severe dementia).
Change in Blessed Dementia Scale score | Baseline, 1-year follow-up, and 2-year follow-up
  This test measures functional deterioration related to dementia. Scores range from 0 (normal function) to 28 (severe dementia-related impairment).
Change in Cardiovascular Risk Factors, Aging, and Incidence of Dementia (CAIDE) score | Baseline, 1-year follow-up, and 2-year follow-up
  CAIDE evaluates long-term dementia risk associated with cardiovascular and lifestyle-related factors. The score is a composite with no fixed scale; a higher score indicates a higher risk.
Change in Cumulative Illness Rating Scale (CRIS) score | Baseline, 1-year follow-up, and 2-year follow-up
  CRIS assesses comorbidity burden across organ systems to quantify illness severity. The score per domain ranges from 0 (no impairment) to 4 (extremely severe), and a summed score is used.
Change in body weight | Baseline, 1-year follow-up, and 2-year follow-up
  Participants' weight is measured to monitor physical health and its association with cognitive and functional outcomes, recorded in kilograms (kg).
Change in body height | Baseline, 1-year follow-up, and 2-year follow-up
  This supports anthropometric analysis by recording participants' height in centimeters (cm).
Change in abdominal circumference | Baseline, 1-year follow-up, and 2-year follow-up
  Measured in cm, this indicates central adiposity and metabolic risk.
Change in blood pressure | Baseline, 1-year follow-up, and 2-year follow-up
  Systolic and diastolic pressures are measured as indicators of cardiovascular health, expressed in millimeters of mercury (mmHg).
Questionnaire for User Interaction Satisfaction (QUIS) | Baseline, 1-year follow-up, and 2-year follow-up
  QUIS evaluates satisfaction with digital tool usability and interaction. Each question is rated from 1 (very poor satisfaction) to 9 (very high satisfaction).
5-level EQ-5D (EQ5D5L) questionnaire | Baseline, 1-year follow-up, and 2-year follow-up
  EQ5D5L measures health-related quality of life across five dimensions. Responses are recorded as five-level categorical options per domain and on a scale from 0 (worst health) to 100 (best imaginable health).
Change in concentration of plasma biomarkers | Baseline, 1-year follow-up, and 2-year follow-up
  Plasma samples are analyzed for phosphorylated tau isoforms (pTau181 and pTau217) to evaluate longitudinal changes related to cognitive decline. Results are reported in picograms per milliliter (pg/mL).
Basal evaluation of CSF biomarkers | Once at the beginning of the study
  CSF samples are analyzed at the beginning of the study for AD biomarkers (amyloid beta 40 (Aβ40) and amyloid beta 42 (Aβ42), phosphorylated tau, total tau), following Alzheimer's Biomarker Standardization Initiative protocols. Units are pg/mL.

OTHER OUTCOMES:
Changes in spontaneous speech evaluation | Every 3-4 months from baseline through 2 years
  The speech assessment involves a picture description task where they describe a given image for one minute, followed by a category fluency task, listing as many items as possible within a given category, such as fruits or professions, within a minute. Finally, open-ended questions prompt participants to describe personal experiences and daily routines. All three tasks are completed within 3 minutes.
Changes in brain MRI | Once at the beginning of the study
  Evaluation of vascular contributions to cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ace Alzheimer Centre Barcelona (Fundació ACE), Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Valero S, Miguel A, Blazquez-Folch J, Calm B, Alegret M, Solivar A, Manias G, Antoniades A, Angelova N, Psimaris D, Segkouli S, Morera A, Tantinya N, Rosende-Roca M, Cano A, Fernandez MV, Sanz-Cartagena P, Gurruchaga MJ, Tarraga L, Boada M, Ruiz A, Marquie M; and COMFORTage Consortium. The COMFORTage project: study protocol for the integration of multiple sources towards personalised preventions at Ace Alzheimer Center Barcelona. Front Digit Health. 2026 Jan 26;7:1633507. doi: 10.3389/fdgth.2025.1633507. eCollection 2025. PMID 41669721